CLINICAL TRIAL: NCT00660361
Title: A Surveillance Program for the Detection of Hepatitis B Virus (HBV) Resistance to Tenofovir (TDF) in HIV-HBV co-Infected Patients
Brief Title: A Surveillance Program for the Detection of Hepatitis B Virus (HBV) Resistance to Tenofovir in HIV-HBV co-Infected Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Bayside Health (Other Government)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Professor Sharon Lewin, The Alfred Hospital and Monash University
Other Study IDs: ALF-50/08
Record Dates: First submitted 2008-04-16; First posted 2008-04-17 (Estimated); Last update posted 2008-04-17 (Estimated); Status verified 2008-04

CONDITIONS: HIV Infections; Hepatitis B Virus
Keywords: HIV; HBV; co-infection; drug resistance; tenofovir; HIV-HBV co-infection
MeSH Terms: conditions — HIV Infections; Hepatitis B; Coinfection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Stored serum samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A: individuals co-infected with HIV-HBV and receiving tenofovir as aprt of their HAART regimen

SUMMARY:
Human immunodeficiency virus/Hepatitis B virus (HIV/HBV) co-infections are frequently observed due to shared routes of transmission, with reported figures indicating 6-9% of HIV-infected individuals in developed countries are chronically infected with HBV. HIV infection impacts on the natural progression of HBV infection, increasing levels of HBV replication and the risk of liver-associated mortality. Liver diseases associated with HBV are affected by the antiviral drugs used for HIV infection (toxic side effects), the current immune function in the patient, by improvements in the immune system brought about by control of the HIV infection, and by the development of resistance to the antiviral agents used for both the hepatitis B and the HIV infection. Tenofovir (TDF) is a newer antiviral drug that is frequently used for HIV infection and is also highly active against hepatitis B; however it is still unknown whether resistance to TDF will eventually develop and how this will affect the long-term outcomes

DETAILED DESCRIPTION:
Tenofovir disoproxil fumarate (TDF) is a nucleotide analogue that can inhibit both HIV and HBV DNA polymerases, and is active against wild-type HBV and HBV strains that contain lamivudine-associated polymerase gene mutations (Dore, Cooper et al. 2004). TDF was approved for use, in combination with other antiretrovirals, for HIV therapy in April 2002 in Australia. It is not currently approved for use in Australia for treatment of HBV mono-infection. TDF has only recently become available in Thailand where HIV/HBV co-infected individuals are predominantly infected with genotype B and C. In contrast, in Australia and Europe, the dominant HBV genotype in HIV/HBV co-infected individuals is A and D. As with all antiviral agents there is concern with long-term use and the development of resistance.

There has been a report of a signature mutation leading to TDF resistance at rtA194T (Sheldon et al., 2005). We recently conducted a retrospective study of HIV/HBV co infected individuals in Melbourne who had received TDF for at least 3 months. Twenty-eight patients had samples available on TDF of which four (~14%) had detectable HBV DNA by PCR. We did not identify the mutation rtA194T or rtV214A/Q215S in individuals failing TDF and found that the only persisting mutations were LMV-resistant mutations. These findings highlight the need for a surveillance system for HIV-HBV co-infected individuals receiving TDF for the detection of novel mutations in the four major HBV genotypes. In addition, it is important to determine the clinical and virological risk factors for TDF failure. This is particularly important given that these agents will be used indefinitely in this patient population and with the development of unique drug resistant mutations there will be implications for progression of liver disease and future therapeutic choices.

This study will recruit patients who are co-infected with HIV and HBV, and are currently taking or who are about to commence the anti-HIV drug TDF. The study cohort will include HIV-HBV co-infected individuals from the Alfred Hospital and Melbourne Sexual Health Clinic. Other sites, not covered by this application, are St Vincent's Hospital, Sydney and King Chulalongkorn Memorial Hospital, Bangkok, Thailand.

The aim of the study is to identify any changes in the HBV DNA that might be associated with resistance to TDF, to determine how long any changes take to occur and to determine the effect of these changes on the clinical response to TDF.

This will be achieved by 6 monthly assessment over a 2 year period, with medical history, physical examination, routine clinical investigations, hepatitis B activity and HBV DNA sequencing.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* HIV positive
* 2 positive Hepatitis B surface antigen results at least 6 months apart
* currently receiving (or about to commence) tenofovir therapy

Exclusion Criteria:

* unable to provide informed consent
* lack of a serum sample prior to commencing tenofovir

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals co-infected with HIV-HBV and currently receiving tenofovir as part of their HAART regimen
Sampling Method: Non-Probability Sample
Enrollment: 92 (Estimated)
Dates: Start 2008-04; Primary Completion 2010-04 (Estimated); Study Completion 2010-09 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Sharon L, MD, PhD, Principal Investigator — The Alfred Hospital and Monash University
Locations (1):
- The Alfred Hospital, Melbourne, Victoria, Australia